CLINICAL TRIAL: NCT01721174
Title: A Randomized Controlled Trial of Endoscopic Biliary Radiofrequency Ablation of Malignant Distal Common Bile Duct Strictures.
Brief Title: Endoscopic Biliary Radiofrequency Ablation of Malignant Distal Common Bile Duct Strictures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2012.153
Record Dates: First submitted 2012-10-31; First posted 2012-11-05 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma
Keywords: Pancreatic cancer; Cholangiocarcinoma; Endoscopic radiofrequency ablation
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEMS only (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the length of the biliary stricture, diameter, and position. An uncovered self expanding metallic stent (SEMS) would be inserted to bypass the site of narrowing (Niti-S biliary uncovered metallic stent; Taewoong Medical, Gimpo City, Korea)
  Interventions: Procedure: SEMS only
- EBRFA and SEMS (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) would be performed under standard operating conditions to confirm the length of the biliary stricture, diameter, and position. The radiofrequency ablation (EBRFA) catheter would be placed under fluoroscopic guidance across the biliary stricture. The Habib EndoHPB (EMcision UK, London, United Kingdom) radiofrequency ablation catheter with energy delivered by an RFA generator would be used to apply RFA to the entire length of the stricture, sequential applications would be applied to complete treatment throughout the length of the stricture without significant overlap of treated areas. Patients would undergo 2 sessions of EBRFA 2 weeks apart. A plastic stent would be inserted in between the 2 sessions. An uncovered SEMSs (Niti-S biliary uncovered metallic stent; Taewoong Medical, Gimpo City, Korea) would be placed after the second EBRFA.
  Interventions: Procedure: EBRFA and SEMS

INTERVENTIONS:
Procedure: SEMS only — The SEMS (Niti-S biliary uncovered metallic stent; Taewoong Medical, Korea) would be placed.
  Arms: SEMS only
Procedure: EBRFA and SEMS — The radiofrequency ablation (RFA) catheter would be placed under fluoroscopic guidance across the biliary stricture. The Habib EndoHPB (EMcision UK, London, United Kingdom) radiofrequency ablation catheter is a bipolar RFA probe that is 8F (2.6 mm), 1.8 m long, compatible with standard (3.2-mm working channel) side-viewing endoscopes, and passes over 0.035-inch guidewires. The catheter has 2 ring electrodes 8 mm apart with the distal electrode 5 mm from the leading edge, providing local coagulative necrosis over a 2.5-cm length. Depending on the length of the stricture, sequential applications would be applied to complete treatment throughout the length of the stricture without significant overlap of treated areas. An uncovered SEMSs (Niti-S biliary uncovered metallic stent; Taewoong Medical, Gimpo City, Korea) would be placed after 2 sessions of EBRFA.
  Arms: EBRFA and SEMS

SUMMARY:
Malignant bile duct obstruction is a common sequela of pancreatic cancers or distal bile duct cancers, and its development can hinder the use of chemotherapy, decrease patient quality of life, and decrease survival. To relieve obstructive jaundice as a result of the obstruction, endoscopic stent placement is usually required. The use self-expandable metal stents (SEMSs) have been shown to result in a longer patency times as compared with plastic stents. However, despite improvements in materials and stent design, stent obstruction still occurs in 13% to 44% of the patients. Tumor in-growth is the most common mechanism of stent obstruction.

Recently, the use of endoscopic biliary radiofrequency ablation (EBRFA) have been described in patients suffering from inoperable malignant distal common bile duct (CBD) obstruction. The procedure uses heat energy to cause local tumour tissue death, resulting in re-opening of the bile duct lumen. The procedure has the potential of reducing the rate of stent obstruction after SEMS and also prolonging survival. The safety profile appears to be comparable that of placement of SEMS alone without added complications (<10%). The aim of the current study is to compare the efficacy of EBRFA with the addition of SEMS to SEMS alone in a randomized controlled trial.We hypothesize that the application of EBRFA can reduce recurrent biliary obstruction after SEMS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old with informed consent
2. Histologically (preferred) or radiologically confirmed distal malignant bile duct tumors
3. Inoperability by staging, comorbidities or patient wishes
4. Distal tumors 2cm away from the portal hilum
5. Bilirubin > 50umol/L at diagnosis

Exclusion Criteria:

1. Periampullary tumours
2. Multiple hepatic metastases with significant blockage of one or more liver segments (if no segment blockage, metastasis is not an exclusion criteria)
3. Presence of main portal vein thrombosis
4. Prior SEMS placement
5. Prior Billroth II or roux-en Y reconstruction
6. History of bleeding disorder or use of anticoagulation
7. Child's B/C cirrhosis
8. Pregnancy
9. Performance status ECOG ≥3 (confined to bed / chair > 50% waking hours)
10. Presence of other malignancy
11. Presence of gastric outlet obstruction
12. Life expectancy < 3months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Stent patency rate | 6 months

SECONDARY OUTCOMES:
Overall survival | 3 years
Serious adverse events | 30 day
Unscheduled readmission rates | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Steel AW, Postgate AJ, Khorsandi S, Nicholls J, Jiao L, Vlavianos P, Habib N, Westaby D. Endoscopically applied radiofrequency ablation appears to be safe in the treatment of malignant biliary obstruction. Gastrointest Endosc. 2011 Jan;73(1):149-53. doi: 10.1016/j.gie.2010.09.031. PMID 21184881